CLINICAL TRIAL: NCT07275385
Title: Advanced Cutaneous Evaluator (ACE): Estimation of Clinical and Economic Impact
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACE
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Wounds and Injuries; Wound Complication
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (non-ACE) (Active Comparator): professionals in the non-ACE group will carry out their usual clinical practice of healing chronic wounds and, in the same way as members of the ACE group, each time they make a decision about local treatment products for these wounds, they must record it in the data collection notebook.
  Interventions: Other: Control (non-ACE)
- ACE (Experimental): The professionals assigned to the ACE group will recruit patients whose wounds will be photographed for use in the application. These images will not be saved but will be deleted immediately after each treatment consultation using the ACE application. Clinical judgment will always prevail. If the professional considers the treatments suggested by ACE unsuitable, they will not apply any of them; instead, they will treat the patient with what they deem best as a healthcare professional. For the purposes of this study, the healthcare professionals in the experimental group will use the software as a clinical decision support system to consult the products they recommend for wound treatment, recommending only wound care products commonly used in participating centers.
  Interventions: Device: Advanced Cutaneous Evaluator (ACE)

INTERVENTIONS:
Device: Advanced Cutaneous Evaluator (ACE) — Nursing staff include the use of ACE in their routine clinical practice to support their chronic wound treatment decision-making process.
  Arms: ACE
Other: Control (non-ACE) — Professionals in the non-ACE group will carry out their usual clinical practice of chronic wound care.
  Arms: control (non-ACE)

SUMMARY:
ACE is a clinical decision support system for selecting appropriate products for the local treatment of chronic wounds. It was designed with a user-centered approach, and its usability and feasibility have been previously validated in pilot studies with nurses. This protocol will allow for the clinical validation of the software in 18 primary care centers, including the quantification of the clinical and economic effects of using the tool over 9 months. It is a mixed-methods design that includes a randomized controlled trial in which nursing staff incorporate the use of ACE into their routine clinical practice to support their decision-making process for chronic wound treatment. It also includes a usability evaluation throughout the study.

DETAILED DESCRIPTION:
To estimate the clinical and economic impact of ACE, wounds will be reviewed at baseline and every two weeks until closure or until the end of the study period. Wound size will be recorded, and whether or not the wound is closed will be noted, with a maximum follow-up period of 16 weeks. A follow-up will be conducted four weeks after wound closure to assess wound dehiscence or other adverse events. Given these wound follow-up periods, only wounds incurred during the first three months of the study, after the completion of professional recruitment and training, will be included for those assigned to the ACE group. A longitudinal study will be conducted in 18 primary care centers in Galicia.

Once the study period is complete, the clinical and economic impact will be evaluated by comparing the following indicators between the two groups: the primary outcome will be wound closure, and secondary outcomes will include wound evolution (including its size every two weeks from the first ulcer assessment and wound bed tissue assessment), length of hospital stay, readmissions, incidence of hospital-acquired injuries, and the cost of products used for wound treatment. Comparative analyses will be performed by subdividing the groups according to the users' experience in chronic wound treatment at the start of the study and according to the type of chronic wound. In addition, instances in which users in the ACE group choose not to follow the application's recommendations will be recorded and quantified.

To evaluate the usability and acceptability of ACE by nursing staff, validated quantitative and standardized tools will be used. Only professionals assigned to the ACE group will participate, using ACE as a decision support tool whenever they need to select products for wound treatment. On one day during the second week of months 2, 4, and 6, the usability and acceptance of the application will be evaluated by the professionals assigned to the ACE group using the System Usability Scale (SUS). Simultaneously, the NASA TLX scale, which quantifies mental workload as an aspect of usability, will be evaluated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals responsible for selecting products for the local treatment of chronic, curable wounds in adult patients.
* Patients with chronic wounds, aged 18 to 100 years.
* Patients with wounds healing by secondary intention, aged 18 to 100 years.
* Patients and/or professionals who have signed the informed consent form for the study.

Exclusion Criteria:

* Minors
* Wounds of patients with acute surgical wounds, aged between 18 and 100 years.
* Images containing features that allow patient identification, such as tattoos and/or moles, or where part of the face is visible.
* Wounds corresponding to third-degree burns, tumor wounds, ischemic ulcers, pyoderma gangrenosum, and ulcers with osteomyelitis without systemic antibiotic treatment.
* Patients and professionals who declined to participate after reading the report Informed Consent Form.

Exclusion criteria:

• During the study, exclusion criteria include wounds lost to follow-up before completing 4 weeks of treatment, except for those that complete follow-up due to wound healing and discharge. Additionally, healthcare professionals and patients who withdraw their consent and wish to leave the study will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Treatment group | Day 0
  ACE or non-ACE
Health center | Day 0
  Open Field
Training of healthcare professionals | Day 0, at the start of the professional's participation
  Academic training of healthcare professionals
Years of experience of healthcare professionals | Day 0, at the start of the professional's participation
  Years of experience of healthcare professionals in healing chronic wounds
SUS | At month 1, month 3 and month 5 after the professional's participation
  Score obtained after completing the System Usability Scale questionnaire
NASA TLX | At month 1, month 3 and month 5 after the professional's participation
  Score obtained after completing the NASA TLX questionnaire
Patient age | Day 0, at the start of recruitment
  Patient's age in years
Gender | Day 0, at the start of recruitment
  Male or female
Diseases | Day 0, at the start of recruitment
  Indicate, if applicable, the following option(s): DM I or II, venous and/or arterial insufficiency, ischemia, obesity, osteomyelitis, diabetic neuropathy, others.
Allergies | Day 0, at the start of recruitment
  Open field
Recurrent medication | Day 0, at the start of recruitment
  Indicate, if applicable, the following option(s): Corticosteroids, NSAIDs, anticoagulants, others.
History of chronic wounds | Day 0, at the start of recruitment
  Indicate, if applicable, etiology, highest classification, location, and if healed, the approximate closing date.
Number of wounds in the same patient | Day 0 and follow-up day every 2 weeks until end of recruitment
  Number
Wound location | Day 0, at the start of recruitment
  Open field
Date of first consultation | Day 0, at the start of recruitment
  Date
Date of wound closure | Day of wound closure after follow-up
  Date
Date of loss to follow-up (if applicable) | Day of loss to follow-up after follow-up
  Date
Reason of loss to follow-up (if applicable) | Day of loss to follow-up after follow-up
  Open field
Date of treatment decision | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Date
Use of ACE? | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Yes or No
Wound size | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Width, length and depth (if applicable) measured in cm
Tissues in the wound bed | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Indicate the following option(s): Necrotic, Sloughing, Granulation, Epithelial, Intact skin with erythema
Dominant tissue in the wound bed | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Select one of the options: Necrotic, Sloughing, Granulation, Epithelial, Intact skin with erythema
Exudate level | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Select one of the options: 0 none, 1 scarce, 2 moderate, 3 abundant
Condition of the perilesional skin | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Indicate the following option(s): Macerated, Erythema or inflammation, Eczema, Fragile skin
Etiology of the wound | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Select one of the options: LESCAH, Diabetic foot, Burn, Arterial, Pressure, Venous, Not determined
Category of the wound | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Indicate the corresponding one according to the selected etiology: LESCAH: 1A/1B/2A/2B; Diabetic foot (Wagner): I/II/III/IV/V; Burn: 1st/2nd/2nd deep/3rd; Arterial: hypertensive ulcer (of Martorell)/arteriosclerotic ulcer/angitic ulcer (of Buerger); Pressure: I/II/III/IV; Venous: C2 (varicose veins)/C3 (edema)/C4a (pigmentation and/or eczema)/C4b (lipodermatosclerosis or white atrophy)/C5 (healed ulceration)/C6 (active ulceration).
Applied products | Day 0 and follow-up day every 2 weeks until wound closure or end of study
  Indicate the following option(s): Actisorb plus 25, Allevyn Adhesive 12, Allevyn Gentle Border 7, Allevyn Heel 13, Allevyn Sacrum 22 x 22 cm, Aquacel Ag, Aquacel Ag + Extra, Aquacel Ag Tape, Aquacel Ag Foam, Aquacel tape, Aquacel Extra, Adhesive Aquacel Foam, Non-Adhesive Aquacel Foam, Aquacel foam pro, Askina carbosorb, Biatain Contact, Biatain non adhesive, Biatain, Silicone with border, Biatain Silicone Without Rim, Cavilon, Comfeel plus sacral, Comfeel plus transparent, Convamax Superabsorb, Conveen Protact, Corpitol, Topical corticosteroid, Cutimed Alginate, Cutimed Sorbact, Cutmed Epiona, Non-sterile Granudacyn, Transparent Hydrotac, Intrasite gel, Iodosorb, Iruxol, Mepilex Border Flex Lite, Mepilex border flex oval, Mepilex border sacrum, Microdacyn 60 Sterile, Trionic, Urgo K2, Urgoclean, Urgoclean AG, Urgostart Plus Pad, Urgotul, Urgotul AG, Varihesive Extra Fine, Varihesive Gel Control, Vliwaktiv AG, Others.
Date of Adverse Event (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Date
Adverse Event classification (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Indicate the following option(s): Severe, Not severe, Expected, Unexpected, Related, Possibly related, Not related
Description of Adverse Event (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Open field describing the event, device deficiency (if applicable), clinical signs, clinical impact, patient action/treatment/outcome.
Measure taken after Adverse Event (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Select one of the options: None, Change of treatment, Other.
Outcome of the Adverse Event (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Select one of the options: Recovered, Recovering, Not recovered, Recovered with sequelae, Fatal, Unknown
Date of resolution of the Adverse Event (if applicable) | Day 0, follow-up day every 2 weeks until wound closure or end of study and 4 weeks after the wound closed
  Date

CONTACTS AND LOCATIONS:
Locations (1):
- Complexo Hospitalario Universitario de Pontevedra, Pontevedra, Spain